CLINICAL TRIAL: NCT06268951
Title: Recovery and Symptom Relief Following Percutaneous Ablation of Abdominal Wall Endometriosis
Status: Enrolling by invitation | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Thomas D. Atwell, Principal Investigator, Mayo Clinic
Other Study IDs: 23-005485
Record Dates: First submitted 2024-02-13; First posted 2024-02-21 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Endometriosis
Keywords: Abdominal Wall endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
To determine the characteristics of recovery and symptom relief following ablation of abdominal wall endometriosis.

DETAILED DESCRIPTION:
The purpose of this study is to characterize the recovery and symptom relief following cryoablation of abdominal wall endometriosis. Patients undergoing clinically indicated ablation of abdominal wall endometriosis will receive an endometriosis-specific symptom survey (Endometriosis Health Profile - 30) prior to ablation and then at 3-, 6-, 12-, and 24-months following treatment. A 2 question survey related to pain at the treatment site will also be administered prior to ablation and then at 1-, 7-, and 30-days after ablation.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing ablation for abdominal wall endometriosis.

Exclusion Criteria:

* Decline to participate in research.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with endometriosis of the abdomen wall.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-05-09 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Symptom severity due to abdominal wall endometriosis following ablation. | Baseline and intermittently over 24 months
  Using the Endometriosis Health Profile - 30 survey, the impact of ablation on endometriosis-related symptoms will be quantified over time. A numerical rating scale will be used to quantify pain at the site of treated abdominal wall endometriosis.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Atwell, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials